CLINICAL TRIAL: NCT04785313
Title: Anatomopathological Analysis and Clinical Evolution After Radiological Removal of Retrievable Vena Cava Filters
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN422021/CHUSTE
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Vena Cava Thrombosis
Keywords: Inferior Vena Cava Filters; Mechanism; Retrievable; Deep Venous Thrombosis; Pathological Evolution; pulmonary embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrievable Inferior Vena Cava Filters (IVCF): The population study includes patients with a Retrievable Inferior Vena Cava Filters (IVCF) placed because of temporary contraindication to curative anticoagulation and that was been removed by the radiology department at the University Hospital of Saint-Etienne, between January 1, 2010 and December 31, 2014. All the Inferior Vena Cava Filters (IVCF) were been sent for histological examination.
  Interventions: Biological: Retrievable Inferior Vena Cava Filters (IVCF); Other: Demographics data collection

INTERVENTIONS:
Biological: Retrievable Inferior Vena Cava Filters (IVCF) — Analysis anatomopathology of Retrievable Inferior Vena Cava Filters (IVCF) (ALN CF model).
Other: Demographics data collection — Demographics data : age, gender, thromboembolic risk factors, Retrievable Inferior Vena Cava Filters (IVCF) (indication, dates of insertion and removal), and anticoagulant management during the period with filter.

SUMMARY:
Pulmonary embolism (PE) is a common pathology causing significant morbidity and mortality. It is usually secondary to migration through the inferior vena cava (IVC) of a formed thrombus in the veins of the lower limbs or pelvis. The inferior vena cava filter (IVCF) is a medical device whose purpose is to prevent thrombus migration from the veins of the legs and pelvis to the pulmonary arteries, thus preventing the occurrence of Pulmonary embolism (PE).

There is no data on the interactions of Retrievable inferior vena cava filters (IVCF) with the inferior vena cava (intrafilter thrombi, insertion through the venous wall) although it may modify the evolution after IVCF retrievable.

DETAILED DESCRIPTION:
The main objective of this study is to determine whether the presence of intrafilter thrombi identified by anatomopathology at the time of inferior vena cava filters (IVCF) retrievable was associated with the occurrence of a venous thromboembolism event within 3 months following removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Inferior Vena Cava Filters (IVCF) placed because of temporary contraindication to curative anticoagulation and that was removed by the radiology department at the University Hospital of Saint-Etienne

Exclusion Criteria:

* Patients included in the PREPIC 2 study
* Patients whose basement filter had not been removed (difficult removal with surgery, no indication for removal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Inferior Vena Cava Filters (IVCF) placed because of temporary contraindication to curative anticoagulation and that was been removed by the radiology department at the University Hospital of Saint-Etienne, between January 1, 2010 and December 31, 2014. All the Inferior Vena Cava Filters (IVCF) were been sent for histological examination.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Correlation between presence of intrafilter thrombi identified by anatomopathologist at the time of retrievable inferior vena cava filters (IVCF) and the occurrence of a venous thromboembolism event within 3 months following removal. | 3 months
  Presence of intrafilter thrombi is measure by anatomopathology analysis of the Inferior Vena Cava Filters (IVCF).
  Venous thromboembolism events are either deep venous thrombosis (DVT) of the lower limbs (diagnosed by Doppler ultrasonography of the lower limbs) or pulmonary embolism (PE) (diagnosed by chest angio-computed tomography).

SECONDARY OUTCOMES:
Correlation between presence of vascular wall fragments and venous thromboembolism event or death within 3 months following removal. | 3 months
  Measured by anatomopathology analysis of the Inferior Vena Cava Filters (IVCF).
Correlation between a high tilt of the Inferior Vena Cava Filters (IVCF) and the occurrence of thromboembolic events within the 3 months following the removal of the Inferior Vena Cava Filters (IVCF) | 3 months
  Tilt was numerically calculated (from 1 to 20) using the Carestream picture archiving communication system (PACS®) for the majority of the patients treated since 2012 and using a protractor on radiological and light boxes films for patients treated 2010 and 2011 (not recorded on the PACS®).
  High Tilt is Tilt > 15.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice-Guy BARRAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No